CLINICAL TRIAL: NCT05200039
Title: Health Status, Quality of Life and Function in Survivors After Radical Treatment for Prostate Cancer. A Cross-sectional Study Focusing on Older Survivors. Part IIB
Brief Title: Health Status, Quality of Life and Function in Survivors After Radical Treatment for Prostate Cancer. Part IIB
Acronym: OPSIIB
Status: Completed | Type: Observational
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 150410-IIB
Record Dates: First submitted 2021-12-16; First posted 2022-01-20 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer; Survivorship; Physical Function; Physical Activity; Old Age
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Older men who were treated for localized or locally advanced prostate cancer with curative intent at the age of 70 years or more
- Matched population based controls: Existing population based data from men who participated in the Trøndelag Health Survey 2017-2019, matched on age and education

SUMMARY:
The present study is the last part of a larger project investigating the health, quality of life and function of men having received radical treatment for prostate cancer in 2014-2018. In this study, physical function and level of physical activity will be tested and registered in a selection of older men who participated in the foregoing parts of the project. Comparisons will be made to similar data from a population-based cohort, matched on age and education.

DETAILED DESCRIPTION:
Background:

Prostate cancer is the most common cancer among Norwegian men with about 5000 new cases each year. Median age at diagnosis is 70 years. Radical treatment for local or locally advanced prostate cancer is either radiotherapy or surgery. Older men more frequently have an aggressive cancer compared to younger men. Despite this, increasing age seems to be a major determinant for omitting curative treatment. Reasons may be worries about side effects in a more vulnerable population, and scarce knowledge about the long-term impact of radical treatment on the older patients' health, function, and quality of life.

Design:

The study is the last part of larger project investigating the health status, quality of life, and function among survivors after radical prostate cancer treatment, focusing on older survivors in particular (NCT04863352). In this study, physical function, physical activity, quality of life, and cardiopulmonary fitness will be evaluated in a subgroup of those men who participated in the foregoing parts of the overarching project, and who were 70 years or more when they received their treatment. The study has a cross-sectional design, and for comparison with a general population, existing data from male participants in the fourth wave of the Trøndelag Health Survey (HUNT4) will be used. The control group will be matched with the study group on age and education, with a distribution 1:3 (cancer survivors : controls).

Aims:

The primary study aim is to investigate if objectively assessed physical performance, physical and sedentary activity in older prostate cancer survivors differ from that of a general male population of the same age.

The secondary aim is to investigate whether and how objectively assessed physical performance is associated with QoL and self-reported physical function and activity.

Study conduct:

To be invited is a random sample of older participants (>70 years old by the time of treatment) in the foregoing parts of the overarching project, stratified by actual age combined with age at treatment. Consenting participants will be invited to testing, which will take place at various hospital locations. The testing will include registration of weight and height, waist circumference, and resting heart rate. Physical performance will be tested by the Short Physical Performance Battery (SPPB), one-legged balance test, and grip strength. Registration of physical- and sedentary activity will be performed using the accelerometer Axivity AX3, which assesses time spent sitting, lying, standing, walking, running, etc. Participants will wear two devices on all waking hours for seven days, one attached to their hip and one to their back. The registrations will be transferred to a designated software for analysis. The participants will also answer a short questionnaire including items on self-reported physical activity and quality of life. Testing is estimated to take about 30-45 min. A PhD student (MD) and a project nurse will perform the testing, instruct the participants how to wear the accelerometers, and to return the devices in a pre-paid envelope. Consenting participants, unable to meet at the arranged occasions, will be tested locally/at home by trained community cancer nurses/physiotherapists.

Statistics:

SPPB scores (primary outcome) will be compared between the older prostate cancer survivors and their matched controls by bivariate linear regression model. Adjustments will be made for potential pre-defined confounders (social status, comorbidity scores, and health status) and matching variables (age and education) to avoid the residual confounding in a multiple linear regression model. Secondary outcomes will be assessed in the same way as the primary ones for each objective. The type of regression model will be considered based on the nature of each outcome analysed.

Sample size: According to Green's rule of thumb, with 10 variables in the multiple model at least 130 participants will be needed to obtain valid estimates. To cover for possible registration failures for some participants, a random sample of 150 consenting older participants who fulfill the inclusion criteria and thrice as many matched controls will be included.

ELIGIBILITY:
Inclusion Criteria, Study group:

* having received radical radiotherapy or robot-assisted radical prostatectomy for prostate cancer at Innlandet Hospital Trust 01.01.2014 and 31.12.2018
* alive and living in Innlandet County
* fluent in Norwegian (orally and in writing)
* provide written informed consent
* age 70 years or more by the time of treatment
* having participated in the foregoing parts of the overarching project, part I and IIA (NCT04863352), both cross-sectional studies using questionnaires/patient reported outcome measures.

Exclusion Criteria:

- survivors with clinically significant relapse (verified metastases/local progression and/or start of lifelong antiandrogen therapy)

Min Age: 70 Years | Sex: Male
Age Groups: Older Adult
Study Population: Study group: Men having received radical treatment for prostate cancer at Innlandet Hospital Trust at the age of 70 years or more, see eligibility criteria
  Control group: For comparison with a general population, a control group of males matched on age and education will be drawn from the Trøndelag Health Survey 4 70+(HUNT4 70+) (2017-2019), which targeted all inhabitants >70 years in Trøndelag County, Norway
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Physical performance | Cross-sectional study, assessment 3 to 7 years afte radical treatment for prostate cancer
  Physical performance as measured by the short physical performance battery (SPPB)

SECONDARY OUTCOMES:
Physical activity | Cross-sectional study, assessment 3 to 7 years afte radical treatment for prostate cancer
  Physical Activity as registered by accelerometer AX3 Axivity
Sedentary activity | Cross-sectional study, assessment 3 to 7 years afte radical treatment for prostate cancer
  Sedentary activity as registered by accelerometer AX3 Axivity
Grip strength | Cross-sectional study, assessment 3 to 7 years afte radical treatment for prostate cancer
  grip strength as measured by dynamometer
one legged balance test | Cross-sectional study, assessment 3 to 7 years afte radical treatment for prostate cancer
  test assessing the participants ability to balance on one leg
cardiorespiratory fitness (CRF) | Cross-sectional study, assessment 3 to 7 years afte radical treatment for prostate cancer
  CRF as estimated from age, gender, BMI/waist circumference, resting heart rate and and physical activity (self-reported, item from the Trøndelag Health Survey)
physical function | Cross-sectional study, assessment 3 to 7 years afte radical treatment for prostate cancer
  physical function as measured by the European Organisation for Research and Treatment of Cancer Quality of life questionnaire - C30 (EORTC QLQ-C30)
global quality of life | Cross-sectional study, assessment 3 to 7 years afte radical treatment for prostate cancer
  global quality of life as measured by the EORTC
self-reported physical activity | Cross-sectional study, assessment 3 to 7 years afte radical treatment for prostate cancer
  self-reported physical activity as measured by items for the Trøndelag Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Marit Slaaen, PhD, Study Chair — Sykehuset Innlandet HF; Ola Berger Christiansen, PhD, Principal Investigator — Sykehuset Innlandet HF
Locations (1):
- Innlandet Hospital Trust, Brumunddal, Norway

IPD SHARING:
Plan to Share IPD: No
According to Norwegian Privacy Protection regulations, data cannot be shared as long as they are not anonymised. However, insight into all data is possible by visiting our research site